CLINICAL TRIAL: NCT04892225
Title: Effect of Text Messages on Dietary Salt and Fluid Restriction on Inter-dialytic Weight Gain in Hemodialysis Patients: A Multicenter Randomized Clinical Trial
Brief Title: Effect of Behavioral Intervention on Interdialytic Weight Gain in Patients Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Farooq Hospital - West Wood Branch (Other)
Responsible Party: Principal Investigator, Dr. Salman Tahir Shafi, Consultant Nephrologist, Farooq Hospital - West Wood Branch
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FHWWMRCT0001
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: End Stage Renal Disease
Keywords: Inter-dialytic weight gain; Fluid and salt restriction; Behavioral intervention; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to text message in Urdu language on dietary sodium and fluid restriction daily for 8 weeks. Control group will not receive any text message.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals in this group will be randomly assigned to text message in Urdu language on dietary sodium and fluid restriction daily for 8 weeks.
  Interventions: Behavioral: Technology-supported behavioral intervention (text message)
- Control group (No Intervention): Randomly assigned Control group will not receive any text message.

INTERVENTIONS:
Behavioral: Technology-supported behavioral intervention (text message) — A simple text message regarding the salt and fluid restriction in order to reduce the inter-dialytic weight gain will be send on daily basis to all the individuals in the intervention group.
  Arms: Intervention group

SUMMARY:
A randomized clinical trial will be conducted in which effect of behavioral intervention (Text message of dietary salt and fluid restriction) on inter-dialytic weight gain in hemodialysis patients. The purpose of this is to evaluate the efficacy of a technology supported intervention for reducing inter-dialytic weight gain and dietary sodium intake in patients undergoing intermittent hemodialysis.

DETAILED DESCRIPTION:
Mortality among hemodialysis (HD) patients remains high with cardiovascular causes accounting for more than one-third of mortality in incident and prevalent end-stage renal disease (ESRD) patients. One factor contributing to poor cardiovascular outcomes is chronic volume overload ,which is a function of excess fluid intake in relation to residual renal function and fluid removal with dialysis treatments. Interdialytic weight gain (IDWG) is an easily measurable parameter in the dialysis unit, routinely assessed at the beginning of the dialysis session. Very few studies have been designed to determine the direct effect of IDWG on morbidity and mortality. Any such effect is confounded by residual renal function and various comorbidities, the effects of which might be difficult to separate from those of IDWG. Most attempts to control IDWG have concentrated on requiring patients to reduce fluid and dietary salt intake. Inter-dialytic weight gain is the result of salt and water intake between 2 hemodialysis sessions. Interdialytic weight gain (IDWG) is commonly used as an indirect measure of fluid intake in HD patients, while considering the daily urine output of the patient. It is used along with clinical symptoms and signs and predialysis blood pressure readings to make decisions regarding the amount of fluid removal during a dialysis session. IDWG is also used as a basis for fluid and salt intake recommendations. High IDWG has detrimental effects on survival, cardiovascular outcomes, and quality of life. A higher IDWG is associated with higher predialysis systolic and diastolic blood pressure ,uncontrolled hypertension which contributes to left ventricular hypertrophy, increasing intradialytic hypotension as a result of higher ultrafiltration rates , and increased morbidity and mortality.

High IDWG is due to poor adherence to fluid restriction and to excessive intake of fluids. Various strategies and interventions have been proposed to control IDWG such as the reduction of dietary salt intake, behavioral interventions aimed at improving the adherence to fluid restriction, the improvement of xerostomia, and the use of lower dialysate sodium concentration. Despite the severe consequences of non-adherence, it has been estimated that 30%-60% of hemodialysis patients do not adhere to a fluid intake guidelines. Various restrictions and barriers such as psychological (low motivation) or social (inadequate support from family, friends), lack of knowledge (lack of understanding of what they were advised), and lack of self-assessment (being unable to judge overall fluid status, fluid intake, or salt consumption) have been shown to be related to failed adherence to fluid restriction strategy. Strategies of behavioral intervention have been used to improve adherence to fluid restriction and to limit IDWG. These strategies aimed to improve motivation, knowledge, social support and education of hemodialysis patients. The behavioral interventions generally used included various approaches, such as behavioral contracting and weekly telephone contacts with patients, patient self-monitoring and behavioral contracting upon adherence, stepped verbal and written reinforcement, group-administered behavioral self-regulation intervention, group education sessions based on trans-theoretical model (states of change), self-efficacy training, and group or individual cognitive behavioral therapy. Numerous randomized controlled studies have been performed, but unfortunately, their results conflict and cannot permit conclusive considerations. It is difficult to compare such studies because of the differences in terms of duration and sample size. Consequently, it is hard to define if certain behavioral interventions are more effective than others. However, what emerges is that the behavioral intervention, although leading to a positive outcome, is temporary and has limited long-term effectiveness. Modest evidence suggests that behavioral intervention strategies (e.g., instruction in self-monitoring, behavioral contracting, and positive reinforcement) may be associated with improved adherence among hemodialysis patients.

The purpose of this behavioral study was to evaluate the efficacy of a technology-supported behavioral intervention (text message) for reducing IDWGs and dietary sodium intake in patients undergoing intermittent HD. The investigators have devised a relatively simplified behavioral intervention(a simple text message regarding fluid and salt restriction) as it will be easier and less cumbersome to perform owing to the educational status and level of understanding of the local population. Moreover, it is less expensive as compared to other interventions and less complicated. Another study which used text message as medium of communication depicted that smoking quit rates for the text messaging intervention group were 36% higher compared to the control group quit rates. Results also suggested that SMS text messaging technology might be a promising way to improve smoking cessation outcomes. This is significant given the relatively wide reach and low cost of text message interventions. Identifying the components that make interventions efficacious will help to increase the effectiveness of such interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age
* Patients with End stage renal disease and on maintenance hemodialysis at least twice a week for at least 1 month
* Patients or immediate family members have access to mobile phones
* Patients are able to read and understand text message in urdu language

Exclusion Criteria:

* Patients with terminal illness and limited life expectancy of less than 1 month
* Patients with Dementia
* Patients with visual impairment
* Patients with Acute Kidney injury requiring hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Mean inter-dialytic weight gain | 8 weeks
  Comparison of mean inter-dialytic weight gain between two groups at the end of 4 week and 8 week period. Average inter-dialytic weight over last week will be used for comparison.

SECONDARY OUTCOMES:
Change in mean inter-dialytic weight gain | 8 weeks
  Comparison of change in mean inter-dialytic weight gain from baseline between two groups at end of 4 week and 8 week period. Average inter-dialytic weight over last week will be used for comparison.
Proportion of patients with high inter-dialytic weight gain | 8 weeks
  Comparison of proportion of patients with high inter-dialytic weight gain (defined as >4% of dry weight) between two groups at end of 4 week and 8 week period. Average inter-dialytic weight over last week will be used for comparison.
Comparison of pre-dialysis systolic and diastolic blood pressure | 8 weeks
  Comparison of Pre-dialysis Systolic and Diastolic Blood Pressure between two groups at end of study of 4 week and 8 week period. Average Pre-dialysis Systolic and Diastolic Blood Pressures over last week will be used for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Farooq Hospital West Wood Branch, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Disentangling the Ultrafiltration Rate-Mortality Association: The Respective Roles of Session Length and Weight Gain — https://cjasn.asnjournals.org/content/8/7/1151.short
- See also: A comparison of attributions, health beliefs, and negative emotions as predictors of fluid adherence in renal dialysis patients: A prospective analysis — https://link.springer.com/article/10.1007/BF02895152
- See also: Differences in Knowledge, Stress, Sensation Seeking, and Locus of Control Linked to Dietary Adherence in Hemodialysis Patients — https://www.frontiersin.org/articles/10.3389/fpsyg.2016.01864/full
- See also: The Relationship Between Social Support and Adherence of Dietary and Fluids Restrictions among Hemodialysis Patients in Iran — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4134167/
- See also: Psychosocial Intervention Improves Depression, Quality of Life, and Fluid Adherence in Hemodialysis — https://jasn.asnjournals.org/content/25/1/196.short